CLINICAL TRIAL: NCT04666883
Title: Aberrant Lympahtic Drainage of Splenic Flexure Cancer: Are Splenic Hilar Nodes Metastases an Underecognized Phenomenon?
Brief Title: Splenic Hilar Nodes in Splenic Flexure Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, Head of Department, University of Rome Tor Vergata
Other Study IDs: REGISTROSPERIMENTAZIONI/21
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Colon Cancer; Metastases, Lymphatic
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Splenic flexure cancer patients: Splenic flexure cancer patients
  Interventions: Other: Review of records and follow up

INTERVENTIONS:
Other: Review of records and follow up — Follow up to identify patients who developed splenic hilar nodal metastases

SUMMARY:
Report the incidence of metastases to the splenic hilar lymphnodes from splenic flexure primaries. This mode of spread has not been previously characterized for these tumours.

ELIGIBILITY:
Inclusion Criteria:

* All splenic flexure cancer patients

Exclusion Criteria:

* No consent to data utilization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer of the splenic flexure of the colon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Splenic hilum nodal metastases | 5 years
  Splenic hilum nodal metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No